CLINICAL TRIAL: NCT03937141
Title: A Phase 2 Efficacy and Safety Trial of ADU-S100 and Pembrolizumab in Adults With Head and Neck Cancer
Brief Title: Efficacy and Safety Trial of ADU-S100 and Pembrolizumab in Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No substantial anti-tumor activity was observed.
Sponsor: Chinook Therapeutics, Inc. (formerly Aduro) (Industry)
Responsible Party: Sponsor
Organization: Chinook Therapeutics, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADU-CL-20
Record Dates: First submitted 2019-04-29; First posted 2019-05-03 (Actual); Results first posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Metastatic Head and Neck Cancer; Recurrent Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — ADU-S100

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ADU-S100 and pembrolizumab (Experimental): All eligible subjects will receive intravenous (IV) infusions of pembrolizumab and intratumoral injections of ADU-S100.
  Interventions: Drug: ADU-S100

INTERVENTIONS:
Drug: ADU-S100 — intratumoral
  Other Names: MIW815

SUMMARY:
ADU-CL-20 is an open-label, multicenter Phase 2 clinical trial to evaluate the efficacy and safety of intratumoral ADU-S100 (also referred to as MIW815) administered with pembrolizumab in the first-line setting. The population will consist of adults with PD-L1 positive recurrent or metastatic HNSCC.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of recurrent or metastatic HNSCC
* Measurable disease as defined by RECIST v1.1
* PD-L1 positive

Exclusion Criteria:

* Diagnosis of recurrent or metastatic carcinoma of the nasopharynx, squamous cell carcinoma of unknown primary histology; or salivary gland or non-squamous histologies (e.g. mucosal melanoma)
* Disease amenable to local therapy with curative intent (surgery or radiation therapy with or without chemotherapy)
* Prior systemic anti-cancer therapy (use of chemotherapeutic agents, targeted small molecules, immunotherapy, or monoclonal antibodies) for the treatment of recurrent or metastatic HNSCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-06-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - University of Arizona Cancer Center, Tucson, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Yale University Cancer Center, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas, Westwood, Kansas
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - University of Maryland, Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Regions Cancer Care Center, Saint Paul, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University Pittsburgh Medical Center Hillman Cancer Center, Pittsburgh, Pennsylvania
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Gogoi H, Mansouri S, Jin L. The Age of Cyclic Dinucleotide Vaccine Adjuvants. Vaccines (Basel). 2020 Aug 13;8(3):453. doi: 10.3390/vaccines8030453. PMID 32823563

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 17 study centers in the United States.
Pre-assignment Details: All enrolled subjects were included in the trial.
Period: Overall Study
Arm/Group | ADU-S100 and Pembrolizumab
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Arm/Group | ADU-S100 and Pembrolizumab
Number analyzed (Participants) | 16
Age, Customized [Count of Participants; unit: Participants]
  < 65 | 12
  >= 65 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Clinical Activity by the Objective Response Rate (ORR; Complete Response [CR] and Partial Response [PR]) Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: To determine ORR of ADU-S100 in combination with pembrolizumab in subjects with recurrent or metastatic head and neck squamous cell cancer (HNSCC). ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1 and as assessed by the investigator.
Time Frame: Up to 25 months
Population: Analysis performed on subjects who had ≥ 1 post-baseline response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | ADU-S100 and Pembrolizumab
Number analyzed (Participants) | 6
Participants
  Complete Response | 1
  Partial Response | 5

ADVERSE EVENTS:
Time Frame: Subjects were followed for serious and non-serious adverse events (AEs) from Screening until 30 days following the last dose of study drug, up to 1 year, 4 months.
Arm/Group | ADU-S100 and Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 6/16
Serious Adverse Events (participants affected / at risk) | 16/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADU-S100 and Pembrolizumab (N=16)
Stress cardiomyopathy (Cardiac disorders) | 1 (1)
Hypophysitis (Endocrine disorders) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) — Acute pancolitis
Localised oedema (General disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Abscess jaw (Infections and infestations) | 1 (1) — Left mandibular abscess
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Bilateral cervical pain
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Scc floor of mouth
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 1 (1) — Left carotid artery restriction
Cerebrovascular accident (Nervous system disorders) | 1 (1) — Stroke
Presyncope (Nervous system disorders) | 1 (1)
Device malfunction (Product Issues) | 1 (1) — G-tube malfunction
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADU-S100 and Pembrolizumab (N=16)
Anaemia (Blood and lymphatic system disorders) | 7 (14)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Aortic valve disease (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (2)
Ear pain (Ear and labyrinth disorders) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypophysitis (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (3)
Eye inflammation (Eye disorders) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (2) — Acute pancolitis
Constipation (Gastrointestinal disorders) | 6 (9)
Diarrhoea (Gastrointestinal disorders) | 8 (10)
Dysphagia (Gastrointestinal disorders) | 3 (4)
Eructation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (2)
Ileus (Gastrointestinal disorders) | 2 (2)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (11)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (7)
Chest pain (General disorders) | 1 (2)
Chills (General disorders) | 5 (8)
Face oedema (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 9 (12)
Hypothermia (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (2)
Injection site discharge (General disorders) | 1 (1)
Injection site pain (General disorders) | 5 (21)
Injection site scab (General disorders) | 1 (1)
Injection site scar (General disorders) | 1 (1)
Injection site swelling (General disorders) | 2 (2)
Injection site vesicles (General disorders) | 1 (1)
Localised oedema (General disorders) | 3 (6)
Oedema peripheral (General disorders) | 2 (2)
Pyrexia (General disorders) | 6 (7)
Secretion discharge (General disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Sarcoidosis (Immune system disorders) | 1 (1)
Abscess jaw (Infections and infestations) | 1 (1)
Candida infection (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 2 (2)
Otitis media (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (3)
Urinary tract infection (Infections and infestations) | 1 (2)
Wound infection (Infections and infestations) | 3 (6)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) — Tracheostomy site bleeding
Procedural pain (Injury, poisoning and procedural complications) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Blood iron decreased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 2 (4)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Platelet count increased (Investigations) | 1 (3)
Weight decreased (Investigations) | 8 (13)
White blood cell count increased (Investigations) | 1 (1)
Decrease appetite (Metabolism and nutrition disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (8)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (7)
Amnesia (Nervous system disorders) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Dysarthria (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (5)
Presyncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Device malfunction (Product Issues) | 1 (1) — G-Tube malfunction
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Complications associated with device (General disorders) | 1 (1) — Abdominal pain, severe, due to feeding tube dislodged
Aphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (2)
Embolism (Vascular disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (2)
Hypotension (Vascular disorders) | 5 (6)
Lymphoedema (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restriction - study results first published in a joint multi-center paper unless (a) no multi-center publication, or (b) ≥18 months has passed since completion of the study. Thereafter, Investigator may publish provided that Investigator: (i) provides a copy of the publication to Chinook ≥ 45 days in advance of submission for publication; (ii) deletes Chinook Confidential Information (other than the Study results) and (iii) submission may be delayed up to 90 days to permit IP filings.

DOCUMENTS (2):
  • Study Protocol (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT03937141/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT03937141/SAP_001.pdf